CLINICAL TRIAL: NCT03828461
Title: Enhancing Evidence-Based Treatment of Hoarding Disorder With Virtual Reality
Brief Title: Hoarding Disorder Treatment With Virtual Reality
Acronym: HDVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Carolyn Rodriguez, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 41899; 1P30AG059307 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Hoarding Disorder; Hoarding; Clutter
Keywords: hoarding disorder; hoarding; clutter
MeSH Terms: conditions — Hoarding Disorder; Hoarding; Speech Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BITS + VR (Experimental): Facilitated group therapy with behavioral practice; 16 weeks
  Interventions: Behavioral: Facilitated group therapy with behavioral practice; 16 weeks

INTERVENTIONS:
Behavioral: Facilitated group therapy with behavioral practice; 16 weeks — Facilitated group therapy for hoarding disorder with behavioral practice

SUMMARY:
This study explores whether a facilitated peer support group called Buried in Treasures (BIT) and a virtual reality decluttering practice can help individuals with clutter challenges.

DETAILED DESCRIPTION:
Individuals with clutter challenges participate in Buried in Treasures Workshop (BIT) that has been shown to improve symptoms of hoarding disorder. The investigators hypothesize that adding virtual reality decluttering practice to the BIT workshop will decrease hoarding symptoms and level of clutter over time.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 55
2. Either gender and all ethno-racial groups
3. Physically healthy male or non-pregnant female.
4. Hoarding Disorder primary condition
5. Willing and able to understand and complete consent and study procedures
6. English speaking
7. Participant should have the technology to host Zoom calls

Exclusion Criteria:

1. Current or past history of bipolar, psychotic or eating disorders, substance dependence, or substance abuse in the last year.
2. Clinically at risk of suicide with Columbia Suicide Severity Rating Scale (C-SSRS) Suicidal Ideation Subscale of 4 or higher (i.e. suicidal intent without specific plan)
3. Major medical or neurological conditions that increase the risk of participation or that would prevent completing assigned behavioral practice tasks.
4. Unable or unwilling to allow study staff into home for home assessment
5. Currently at high risk for eviction
6. Animal hoarding or squalor

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn I Rodriguez, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Psychiatry Department, Stanford, California, United States

REFERENCES:
- [Background] Raila H, Avanesyan T, Valentine KE, Koo B, Huang C, Tsutsumi Y, Andreeff E, Qiu T, Munoz Rodriguez PA, Varias A, Filippou-Frye M, van Roessel P, Bullock K, Periyakoil VS, Rodriguez CI. Augmenting group hoarding disorder treatment with virtual reality discarding: A pilot study in older adults. J Psychiatr Res. 2023 Oct;166:25-31. doi: 10.1016/j.jpsychires.2023.08.002. Epub 2023 Aug 9. PMID 37716272
- See also: Rodriguez Lab Website — http://med.stanford.edu/rodriguezlab.html
- See also: Dr. Carolyn Rodriguez Faculty Page — https://med.stanford.edu/profiles/carolyn-rodriguez?tab=bio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BITS + VR
Started | 13
Completed | 9
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | BITS + VR
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Hoarding Symptom Severity as Measured by Saving Inventory-Revised (SI-R)
Description: The Saving Inventory-Revised scale (SI-R) is a 23-item questionnaire with 3 factor-analytically defined sub-scales for difficulty discarding, excessive clutter, and compulsive acquisition.
  The total score (sum of 23 items) ranges from 0 to 92. Total score higher than 41 shows significant difficulty with clutter.
  For the acquisition subscale we sum items 2 (reverse score), 9, 11, 14, 16, 18 and 21. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with excessive acquisition.
  For the difficulty discarding subscale we sum items 4(reverse score), 6, 7, 13, 17, 19, 23. The subscale ranges from 0 to 28 and score greater than 13 indicates difficulty with discarding.
  For the clutter subscale we sum items 1, 3, 5, 8, 10, 12, 15, 20, 22. The subscale ranges from 0 to 36 and score greater than 15 indicates difficulty with accumulated clutter.
Time Frame: Change from baseline to 16 weeks after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BITS + VR
Number analyzed (Participants) | 9
score on a scale | 14.2 (7.7)

2. Secondary Outcome: Change in the Severity of Clutter Level as Measured by Clutter Image Rating Scale
Description: Clutter Imaging Rating (CIR) Scale consists of three sets of photographs of a room, each containing nine photos with varying levels of clutter. This scale assesses the clutter levels in the bedroom, living room and kitchen. Patients were asked to select the picture "that most accurately reflects the amount of clutter in your room". Scores on range from 1 (least cluttered) to 9 (most cluttered). A mean composite score ranging from 1 to 9 was calculated across the three rooms for each individual. A cut-off score of 4 or higher indicate significant clutter.
Time Frame: Change from baseline to 16 weeks after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | BITS + VR
Number analyzed (Participants) | 9
score on a scale | 0.77 (0.58)

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Arm/Group | BITS + VR
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BITS + VR (N=9)
dizziness (Nervous system disorders) | 3 (3) — dizziness
general discomfort (Nervous system disorders) | 7 (7)
fatigue (Nervous system disorders) | 3 (3)
headache (Nervous system disorders) | 3 (3)
eye strain (Eye disorders) | 5 (5)
difficulty focusing (Eye disorders) | 5 (5)
salivation increasing (Gastrointestinal disorders) | 1 (1)
sweating (Skin and subcutaneous tissue disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
difficulty concentrating (Nervous system disorders) | 2 (2)
fullness of head (Nervous system disorders) | 3 (3)
blurred vision (Eye disorders) | 4 (4)
veritgo (Nervous system disorders) | 3 (3)
stomach awareness (Gastrointestinal disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03828461/Prot_SAP_000.pdf